CLINICAL TRIAL: NCT02552550
Title: Analysis of Swallowing, Speech and Quality of Life of Patients With Stage T3-T4 Squamous Cell Carcinoma of the Oropharynx Before and After Multimodal Treatment With Curative Intent
Brief Title: Swallowing, Speech and Quality of Life of Patients With Carcinoma of the Oropharynx
Status: Terminated | Type: Observational
Why Stopped: rate of inclusion too low
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1208112; 2012-A00904-39 (Other: ANSM)
Record Dates: First submitted 2015-09-11; First posted 2015-09-17 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
Keywords: squamous cell carcinoma of the oropharynx; swallowing, speech; quality of life
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Speech | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ability to swallow, speak and quality of life: This will just be an evaluation, before any treatment, his ability to swallow, speak and quality of life then, as in normal practice, after 3, 6 and 12 months after treatment.
  Interventions: Procedure: Ability to swallow, speak and quality of life

INTERVENTIONS:
Procedure: Ability to swallow, speak and quality of life — This study will not change the patient's treatment. This will just be an evaluation, before any treatment, his ability to swallow, speak, then his quality of life, as in normal practice, after 3, 6 and 12 months after treatment.

SUMMARY:
The curative treatment and organ preservation in advanced squamous cell carcinoma of the oropharynx is multimodal. It involves induction chemotherapy and depending on the response radio-chemotherapy or surgery. The combination of these methods has important functional consequences.

The aim of this prospective pilot study is to describe swallowing, speech, but also patients' quality of life before and after therapeutic management (existing studies measuring these functions after treatment but not before).

DETAILED DESCRIPTION:
This study will not change the patient's treatment. This will just be an evaluation, before any treatment, his ability to swallow, speak then, as in normal practice, after 3, 6 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stage T3 or T4 squamous cell carcinoma of the oropharynx previously untreated.
* Performance status 0 or 1
* Tumor histology proving squamous cell carcinoma

Exclusion Criteria:

* Visceral metastases at initial assessment
* Contraindication to surgery and / or chemotherapy such as:
* A history of other cancer (except basal cell carcinoma skin or cervical cancer in situ)
* 2nd associated cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patietn with T3 or T4 stage squamous cell cancer of the oropharynx
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-07-25 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

PRIMARY OUTCOMES:
change from swallowing disorder | between day 0 and 1 year
  A swallowing disorder will be determined by conducting a video-endoscopy and voluntary swallowing reflex (composite measure)

SECONDARY OUTCOMES:
Change from phonation disorder | between day 0 and 1 year
  Phonation disorders will be evaluated by the scale "Voice Handicap Index" (composite measure)
Change from quality of life | between day 0 and 1 year
  The quality of life will be assessed by the Quality of Life scale EORTC QLQ-C30 and QLC-HN35 (composite measure)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel PRADES, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHu de SAINT-ETIENNE, Saint-Etienne, France